Official Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study of

Atezolizumab Plus Carboplatin and Etoposide With or Without Tiragolumab in Patients with Untreated Extensive-Stage Small Cell

Lung Cancer

NCT Number: NCT04665856

**Document Date:** Statistical Analysis Plan Version 1: 27-May-2022

#### STATISTICAL ANALYSIS PLAN

STUDY A PHASE III, RANDOMIZED, DOUBLE-BLIND,

TITLE: PLACEBO-CONTROLLED STUDY OF ATEZOLIZUMAB PLUS

CARBOPLATIN AND ETOPOSIDE WITH OR WITHOUT TIRAGOLUMAB IN PATIENTS WITH UNTREATED EXTENSIVE-STAGE SMALL CELL LUNG CANCER

STUDY NUMBER: YO42373

STUDY NAME: SKYSCRAPER-02C

VERSION NUMBER: 1

**ROCHE COMPOUND(S):** Tiragolumab (RO7092284)

Atezolizumab (RO5541267)

**EUDRACT NUMBER:** Not applicable

**IND NUMBER:** 129258

NCT NUMBER: NCT04665856

PLAN PREPARED BY: , Ph.D.

| STATISTICAL ANALYSIS PLAN APPROVAL | |
|---|---|
| SPONSOR:<br>LEGAL REGISTERED<br>ADDRESS: | F. Hoffmann-La Roche Ltd<br>Grenzacherstrasse 124<br>4070 Basel, Switzerland |
| DATE FINAL: | See electronic date stamp on the last page of this document |

#### CONFIDENTIAL

This is an F. Hoffmann-La Roche Ltd document that contains confidential information. Nothing herein is to be disclosed without written consent from F. Hoffmann-La Roche Ltd.

# STATISTICAL ANALYSIS PLAN VERSION HISTORY

| SAP Version | Approval Date | Based on Protocol<br>(Version, Approval Date) |
|---|---|---|
| 1 | see electronic date stamp<br>on the last page of this<br>document | Version 4, 7 October 2021 |

# **TABLE OF CONTENTS**

| 1. | | INTRODUCTION | 8 |
|---|---|---|---|
| | 1.1 | Objectives and Endpoints and Estimands | 8 |
| | 1.1.1 | Expression of Objectives and Endpoint using the Estimand Framework | 11 |
| | 1.2 | Study Design | 14 |
| | 1.2.1 | Treatment Assignment and Blinding | 16 |
| | 1.2.2 | Data Monitoring | 17 |
| 2. | | STATISTICAL HYPOTHESES | 17 |
| 3. | | SAMPLE SIZE DETERMINATION | 18 |
| | 3.1 | Co-Primary Endpoint: Progression-Free Survival in the Primary Analysis Set | 18 |
| | 3.2 | Co-Primary Endpoint: Overall Survival in the Primary Analysis Set | 18 |
| 4. | | ANALYSIS SETS | 19 |
| 5. | | STATISTICAL ANALYSES | 20 |
| | 5.1 | General Consideration | 20 |
| | 5.2 | Patient Disposition | 20 |
| | 5.3 | Primary Endpoints Analysis | <mark>2</mark> 0 |
| | 5.3.1 | Definition of Co-Primary Endpoints | <mark>2</mark> 0 |
| | 5.3.1.1 | Progression-Free Survival | <mark>2</mark> 0 |
| | 5.3.1.2 | Overall Survival | 21 |
| | 5.3.2 | Main Analytical Approach for Primary Endpoints | 22 |
| | 5.3.3 | Handling of Missing Data | 22 |
| | 5.3.4 | Sensitivity Analyses for Primary Endpoints | 22 |
| | 5.3.5 | Supplementary Analyses for Primary Endpoints | 22 |
| | 5.3.5.1 | Subgroup Analyses for Primary Endpoints | 22 |
| | 5.4 | Secondary Endpoints Analyses | 23 |
| | 5.4.1 | Key Secondary Endpoints | 23 |
| | 5.4.1.1 | Progression-Free Survival and Overall Survival in the Full Analysis Set | 23 |
| | 5.4.1.2 | Confirmed Overall Response Rate | 23 |

| Supportive Secondary Endpoint(s) | 24 |
|---|---|
| Duration of Response | 24 |
| PFS and OS Rates at Selected Time Points | 24 |
| Time to Confirmed Deterioration in Physical Functioning and Global Health Status | 24 |
| Exploratory Endpoints Analysis | 26 |
| Patient Reported Outcomes | 26 |
| Biomarker Analyses | 26 |
| Safety Analyses | 27 |
| Extent of Exposure | 27 |
| Adverse Events | 27 |
| Laboratory Data | 28 |
| Vital Signs | 28 |
| Other Analyses | 28 |
| Summaries of Conduct of Study | 28 |
| Summaries of Treatment Group Comparability | 28 |
| Pharmacokinetic Analyses | 28 |
| Immunogenicity Analyses | 28 |
| Interim Analyses | <b>2</b> 9 |
| Planned Interim Analyses | 29 |
| SUPPORTING DOCUMENTATION | 29 |
| REFERENCES | 29 |
| LIST OF TABLES | |
| Objectives and Estimands | 12 |
| | 18 |
| | 10 |
| Analysis Sets | 19<br>19 |
| | and Global Health Status Exploratory Endpoints Analysis Patient Reported Outcomes Biomarker Analyses Safety Analyses Extent of Exposure Adverse Events Laboratory Data Vital Signs Other Analyses Summaries of Conduct of Study Summaries of Treatment Group Comparability Pharmacokinetic Analyses Immunogenicity Analyses Interim Analyses Planned Interim Analyses SUPPORTING DOCUMENTATION REFERENCES Dijectives and Corresponding Endpoints Objectives and Estimands |

# **LIST OF FIGURES**

| Figure 1 Study Schema | 1 | 5 |
|-----------------------|---|---|
|-----------------------|---|---|

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation or Term | Description |
|---|---|
| ACE | atezolizumab and carboplatin and etoposide |
| ADA | anti-drug antibody |
| AE | adverse event |
| AESI | adverse event of special interest |
| ASTCT | American Society for Transplantation and Cellular Therapy |
| CE | carboplatin and etoposide |
| CI | confidence interval |
| CR | complete response |
| CRS | cytokine-release syndrome |
| CSR | Clinical Study Report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DOR | duration of response |
| ECOG | Eastern Cooperative Oncology Group |
| EC | Ethics Committee |
| EORTC | European Organization for the Research and Treatment of Cancer |
| ES-SCLC | extensive-stage small cell lung cancer |
| FAS | full analysis set |
| GHS | global health status |
| HR | hazard ratio |
| ICH | International Council on Harmonization |
| iDMC | independent Data Monitoring Committee |
| iDCC | independent Data Coordinating Center |
| IL46 | item list 46 |
| IRB | Institutional Review Board |
| IRF | Independent Review Facility |
| ITT | intent to treat |
| IxRS | interactive voice/web-based response system |
| LDH | lactate dehydrogenase |
| MDD | minimally detectable difference |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NCI | National Cancer Institute |
| NPT | non-protocol anti-cancer therapy |
| ORR | overall response rate |
| OS | overall survival |

| Abbreviation or Term | Description |
|----------------------|------------------------------------------------|
| PAS | primary analysis set |
| Pbo | placebo |
| PFS | progression-free survival |
| PK | pharmacokinetic |
| PR | partial response |
| PRO | patient-reported outcomes |
| QLQ-C30 | Quality-of-Life Questionnaire Core 30 |
| QoL | Quality of Life |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| RPSFT | Rank-preserving structural failure time |
| SAE | serious adverse events |
| SAP | Statistical Analysis Plan |
| SMQs | standardized MedDRA queries |
| TIGIT | T-cell immunoreceptor with Ig and ITIM domains |
| TTCD | time to confirmed deterioration |
| Tira | tiragolumab |
| ULN | upper limit of normal |

# 1. INTRODUCTION

This Statistical Analysis Plan (SAP) provides details of the planned analyses and statistical methods for Study YO42373 (SKYSCRAPER-02C), a Phase III, randomized, double-blind, placebo-controlled study of atezolizumab plus carboplatin and etoposide (CE) with or without tiragolumab (anti- T-cell immunoreceptor with Ig and ITIM domains [TIGIT] antibody) in Chinese patients with untreated extensive-stage small cell lung cancer (ES-SCLC). The background for the study can be found in the study protocol.

#### 1.1 OBJECTIVES AND ENDPOINTS AND ESTIMANDS

Study YO42373 evaluates the efficacy, safety, and pharmacokinetics (PK) of tiragolumab plus atezolizumab and CE (hereinafter referred to as Tira+ACE) compared with placebo plus atezolizumab and CE (hereinafter referred to as Pbo+ACE) in patients with untreated ES-SCLC. Specific objectives and corresponding endpoints for the study are outlined in Table 1.

The term "study treatment" refers to all protocol-mandated treatments assigned to patients as part of this study and includes Tira+ACE or Pbo+ACE during the induction phase; tiragolumab/placebo and atezolizumab during the maintenance phase.

Table 1 Objectives and Corresponding Endpoints

| Primary Objective(s) | Corresponding Endpoint(s) |
|---|---|
| To evaluate the efficacy of tiragolumab plus atezolizumab and CE compared with placebo plus atezolizumab and CE in patients with previously untreated ES-SCLC without presence or history of brain metastases at baseline (defined as PAS, see Section 4) | <ul> <li>PFS: defined as the time from randomization to the first occurrence of disease progression as determined by the investigator according to RECIST v1.1 or death from any cause, whichever occurs first</li> <li>OS: defined as the time from randomization to death from any cause</li> </ul> |

 Table 1
 Objectives and Corresponding Endpoints (cont.)

| Secondary Objective(s) | Corresponding Endpoints |
|---|---|
| To evaluate the efficacy of tiragolumab plus atezolizumab and CE compared with placebo plus atezolizumab and CE | <ul> <li>PFS in patients with untreated ES-SCLC (defined as FAS, see Section 4)</li> <li>OS in the FAS</li> <li>Confirmed ORR: defined as the proportion of patients with a confirmed objective response (i.e., CR or PR on two consecutive occasions ≥4 weeks apart), as determined by the investigator according to RECIST v1.1 in patients with measurable disease at baseline</li> </ul> |
| | DOR for patients with confirmed objective response, defined as the time from the first occurrence of a documented, confirmed objective response to disease progression, as determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurs first |
| | PFS rates at 6 months and at 12 months, defined as the proportion of patients who have not experienced disease progression as determined by the investigator according to RECIST v1.1 or death from any cause at 6 months and 12 months after randomization |
| | OS rates at 12 months and at 24 months,<br>defined as the proportion of patients who<br>have not experienced death from any cause<br>at 12 months and 24 months after<br>randomization |
| To evaluate the safety of<br>tiragolumab plus atezolizumab<br>and CE compared with placebo<br>plus atezolizumab and CE | Incidence and severity of adverse events, with severity determined according to NCI CTCAE, v 5.0 Severity for CRS will also be determined according to the ASTCT CRS consensus grading scale |

Table 1 Objectives and Corresponding Endpoints (cont.)

| Secondary Objective(s) | Corresponding Endpoints |
|---|---|
| To characterize the tiragolumab and atezolizumab PK profile | Serum concentrations of tiragolumab and atezolizumab at specified timepoints |
| To evaluate the immune response to tiragolumab | <ul> <li>Prevalence of ADAs to tiragolumab at<br/>baseline and incidence of ADAs to<br/>tiragolumab during the study</li> </ul> |
| To evaluate the quality of life of patients treated with tiragolumab plus atezolizumab and CE compared with placebo plus atezolizumab and CE | <ul> <li>TTCD in patient-reported physical<br/>functioning and GHS/QoL, as measured by<br/>the EORTC QLQ-C30</li> </ul> |
| Exploratory Objective(s) | Corresponding Endpoints |
| • | |
| • | |

## Table 1 Objectives and Corresponding Endpoints (cont.)

ADA=anti-drug antibody; ASTCT=American Society for Transplantation and Cellular Therapy; CE= carboplatin and etoposide; CTCAE=Common Terminology Criteria for Adverse Events; CR=complete response; CRS=cytokine-release syndrome; DOR=duration of response; EORTC=European Organisation for the Research and Treatment of Cancer; ES-SCLC=extensive-stage small cell lung cancer; FAS=full analysis set; GHS=Global Health Status; NCI=National Cancer Institute; ORR=objective response rate; OS=overall survival; PAS=primary analysis set; PFS=progression-free survival; PR=partial response; PK=pharmacokinetic; QLQ-C30=Quality-of-Life Questionnaire Core 30; RECIST=Response Evaluation Criteria in Solid Tumors; TTCD=Time to confirmed deterioration.

# 1.1.1 <u>Expression of Objectives and Endpoint using the Estimand</u> Framework

Primary endpoints and key secondary endpoints are expressed using the estimand framework in Table 2, following the International Conference on Harmonization E9 (R1) statistical principles for clinical trials (ICH 2020).

Table 2 Objectives and Estimands

| Primary Objective(s) | Estimand Definition |
|---|---|
| To evaluate the efficacy of tiragolumab plus atezolizumab and CE compared with placebo plus atezolizumab and CE in patients with previously untreated ES-SCLC without presence or history of brain | Population: Patients with previously untreated ES-SCLC without presence or history of brain metastases at baseline |
| | <ul> <li><u>Variable</u>: Time from randomization to the<br/>first occurrence of the respective event of<br/>interest (as defined in <u>Table 1</u>).</li> </ul> |
| metastases at baseline | • <u>Treatments:</u> |
| | <ul> <li>Experimental:<br/>tiragolumab+ atezolizumab+ CE<br/>(induction phase; four 21-day cycles)<br/>followed by tiragolumab+ atezolizumab<br/>(maintenance phase; 21-day cycles)</li> </ul> |
| | <ul> <li>Control: placebo+ atezolizumab+ CE (induction phase; four 21-day cycles) followed by placebo+atezolizumab (maintenance phase; 21-day cycles)</li> </ul> |
| | • Intercurrent events: |
| | <ul> <li>Start of NPT prior to the respective event<br/>of interest</li> </ul> |
| | <ul> <li>Early discontinuation from study<br/>treatment for any reason prior to the<br/>respective event of interest</li> </ul> |
| | Handling of intercurrent events: A treatment-policy with regards to the intercurrent events listed above will be applied for the primary analysis |
| | Summary measure: Hazard ratio for the |

respective variable

Table 2 Objectives and Estimands (cont.)

| Selected Secondary Objective(s) | Estimand Definition |
|---|---|
| Evaluate the efficacy of tiragolumab plus atezolizumab and CE compared with placebo | The estimands for OS and PFS as secondary endpoints are defined similarly as for the primary endpoints except the following: |
| plus atezolizumab and CE | Population: Patients with previously untreated ES-SCLC |
| | The estimand for secondary endpoint of confirmed ORR is defined similarly as for the primary endpoints in terms of population and treatments; the other attributes are defined as follows: |
| | • <u>Variable</u> : |
| | <ul> <li>Whether patients achieved a confirmed<br/>objective response (i.e., CR or PR on two<br/>consecutive occasions ≥4 weeks apart),<br/>as determined by the investigator<br/>according to RECIST v1.1</li> </ul> |
| | Intercurrent events: |
| | <ul> <li>Start of NPT prior to the variable of<br/>interest is observed</li> </ul> |
| | <ul> <li>Early discontinuation from study<br/>treatment for any reason prior to the<br/>variable of interest is observed</li> </ul> |
| | Handling of intercurrent events: A treatment-<br>policy with regards to the intercurrent events<br>listed above will be applied for the analysis<br>of confirmed ORR |
| | Summary measure: |
| | Difference in proportions |

# Table 2 Objectives and Estimands (cont.)

 To evaluate the quality of life of patients treated with tiragolumab plus atezolizumab and CE compared with placebo plus atezolizumab and CE The estimand for secondary endpoint of TTCD is defined similarly as for the primary endpoints in terms of population and treatments; the other attributes are defined as follows:

- Variable: Time from randomization until the first confirmed clinically meaningful deterioration on physical functioning and GHS/QoL using the EORTC QLQ-C30 select scales; confirmed clinically meaningful deterioration is defined as a clinically meaningful decrease from baseline that must be held for at least two consecutive assessments or an initial clinically meaningful decrease from baseline followed by death from any cause within 3 weeks.
- Intercurrent events:
  - Start of NPT prior to a confirmed clinical meaningful deterioration
  - Early discontinuation from study treatment for any reason prior to a confirmed clinical meaningful deterioration
  - Death that occurs before patients report any clinically meaningful deterioration
- Handling of intercurrent events: A treatment policy strategy with regards to the start of NPT and early discontinuation; and whileon-treatment/while-alive strategy for death will be applied for the TTCD analysis.
- Summary measure: Hazard Ratio for TTCD

CE=carboplatin and etoposide; CR=complete response; ES-SCLC=extensive-stage small cell lung cancer; EORTC=European Organization for Research and Treatment of Cancer; GHS=global health status; NPT=non-protocol anti-cancer therapy; ORR=objective response rate; OS=overall survival; PFS=progression-free survival; PR=partial response; QLQ-C30=Quality-of-Life Questionnaire Core 30; TTCD=time to confirmed deterioration.

#### 1.2 STUDY DESIGN

This is a Phase III, randomized, double-blind, placebo-controlled multicenter study in China designed to evaluate the safety and efficacy of tiragolumab plus atezolizumab and CE compared with placebo plus atezolizumab and CE in patients with chemotherapy-naive ES-SCLC.

Eligible patients are stratified by Eastern Cooperative Oncology Group (ECOG) Performance Status (0 vs. 1) and lactate dehydrogenase (LDH) (≤upper limit of normal [ULN] vs.> ULN), and will be randomized 1:1 to receive one of the following treatment regimens:

- Arm A: tiragolumab + atezolizumab + CE (induction phase; four 21-day cycles)
   followed by tiragolumab + atezolizumab (maintenance phase; 21-day cycles)
- Arm B: placebo+ atezolizumab+CE (induction phase; four 21-day cycles) followed by placebo+ atezolizumab (maintenance phase; 21-day cycles)

The study schema is shown in Figure 1.

Figure 1 Study Schema



CE=carboplatin and etoposide; ECOG PS=Eastern Cooperative Oncology Group performance scale; ES-SCLC= extensive-stage small cell lung cancer; FAS=full analysis set; LDH=lactate dehydrogenase; n=number of patients; PAS= primary analysis set; RECIST=Response Evaluation Criteria in Solid Tumors; ULN=upper limit of normal.

Following the induction phase, patients will continue maintenance therapy with either tiragolumab plus atezolizumab (Arm A) or placebo plus atezolizumab (Arm B).

Treatment will be continued until radiographic disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, or as long as patients are experiencing clinical benefit, as assessed by the investigator, in the absence of unacceptable toxicity or symptomatic deterioration attributed to disease progression after an integrated assessment of radiographic data, biopsy results (if available), and clinical status. Patients who meet the criteria for disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 will be permitted to continue study treatment (atezolizumab plus tiragolumab or atezolizumab plus placebo) if they meet all of the criteria specified in study protocol (see Protocol, Section 3.1.2) and provide written consent.

Patients will undergo tumor assessments at baseline and every 6 weeks (±7 days) for 48 weeks following Cycle 1, Day 1, regardless of treatment dose delays. After completion of the Week 48 tumor assessment, tumor assessments will be required every 9 weeks (±7 days) thereafter, regardless of treatment dose delays. Patients will undergo tumor assessments until radiographic disease progression per RECIST v1.1, withdrawal of consent, study termination by the Sponsor, or death, whichever occurs first. Patients who are treated beyond disease progression per RECIST v1.1 will undergo tumor assessments at the frequency described above until study treatment is discontinued. Patients who discontinue treatment for reasons other than radiographic disease progression per RECIST v1.1 (e.g., toxicity, symptomatic deterioration) will continue scheduled tumor assessments at the frequency described above until radiographic disease progression per RECIST v1.1, withdrawal of consent, study termination by the Sponsor, or death, whichever occurs first), regardless of whether the patient starts a new anti-cancer therapy.

### 1.2.1 Treatment Assignment and Blinding

This is a Phase III, randomized, double-blind, placebo-controlled multicenter study. After written informed consent has been obtained and eligibility has been established, the study site will obtain the patient's identification number and treatment assignment from the interactive voice or web-based response system (IxRS).

Patients will be randomized to one of two treatment arms:

- Arm A: tiragolumab + atezolizumab + CE
- Arm B: placebo+atezolizumab+CE

Randomization will occur in a 1:1 ratio through use of a permuted-block randomization method to ensure that an approximately equal number of patients will be enrolled in

each treatment arm within the baseline characteristics of the following stratification factors:

- ECOG Performance Status (0 vs. 1)
- LDH (≤ ULN vs. > ULN)

Patients should receive their first dose of study drug on the day of randomization if possible. If this is not possible, the first dose should occur within 5 days after randomization.

Study site personnel (with the exception of the unblinded pharmacist) and patients will be blinded to treatment assignment during the study. The Sponsor and its agents will also be blinded to treatment assignment, with the exception of individuals who require access to patient treatment assignments to fulfill their job roles during a clinical trial. These roles include the unblinding group responsible, clinical supply chain managers, sample handling staff, operational assay group personnel, IxRS service provider, and Independent Data Monitoring Committee (iDMC) members.

# 1.2.2 <u>Data Monitoring</u>

An iDMC will be used to evaluate safety during the study. The safety review of unblinded data by the iDMC will occur approximately every 6 months. The safety data will include disposition, demographic data, adverse events, serious adverse events, and relevant laboratory data.

The Sponsor will remain blinded to the efficacy results until the primary progression-free survival (PFS) analysis. All summaries and analyses by treatment arm for the iDMC reviews will be prepared by an external independent Data Coordinating Center (iDCC). Following the data review, the iDMC will provide a recommendation as to whether the study may continue, whether amendment(s) to the protocol should be implemented, or whether the study should be stopped. The final decision will rest with the Sponsor, taking into consideration the iDMC's recommendation.

Members of the iDMC will be external to the Sponsor and will follow a separate iDMC Charter that outlines their roles and responsibilities, as well as a detailed monitoring plan.

Any outcomes of these safety reviews that affect study conduct will be communicated in a timely manner to the investigators for notification of the sites' Institutional Review Boards/Ethics Committees (IRBs/ECs).

#### 2. STATISTICAL HYPOTHESES

The emphasis of efficacy analyses is to assess whether the treatment benefit in Chinese patients is consistent with the results observed in the global GO41767 study. The study is not powered to demonstrate statistical significance in terms of efficacy, and no formal

hypothesis testing will be performed. Thus, the hypothesis testing is considered exploratory in this bridging study.

#### 3. <u>SAMPLE SIZE DETERMINATION</u>

Approximately 128 patients, including approximately patients without presence or history of brain metastases at baseline, are planned for enrollment.

# 3.1 Co-Primary Endpoint: Progression-Free Survival in the Primary Analysis Set

The primary analysis of the co-primary endpoint of PFS will be conducted at the time of the OS primary analysis. The analyses are expected to occur at approximately months after the first patient is randomly assigned, with the assumptions on accrual over a period of approximately 13 months. At the time of the primary analysis of PFS, it is estimated that approximately PFS events (PFS) will be determined at the time of OS primary analysis.



- PFS curve following one-piece exponential distributions
- Median PFS of months in Arm A and months Arm B, corresponding to a target hazard ratio (HR) of
- Dropout rate of over 12 months for PFS



# 3.2 Co-Primary Endpoint: Overall Survival in the Primary Analysis Set

- OS curve following one-piece exponential distributions
- Median OS of months for Arm A and months for Arm B, corresponding to a target HR of
- Dropout rate of over 24 months for OS





# 4. ANALYSIS SETS

The analysis sets used for the analyses are defined in the Table 5 below:

Table 5 Analysis Sets

| Analysis set | Definition |
|---|---|
| Full analysis set (FAS) | All randomized patients, whether or not the patient received the assigned treatment |
| Primary analysis set (PAS) | All randomized patients without presence or history of brain metastases at baseline |
| Safety evaluable set | All randomized patients who received at least one dose of study treatment |
| Atezolizumab<br>PK-evaluable set | All patients who received at least one dose of atezolizumab treatment and who have at least one post-baseline PK sample available |
| Tiragolumab<br>PK-evaluable set | All patients who received at least one dose of tiragolumab treatment and who have at least one post-baseline PK sample available |

ADA = anti-drug antibody; FAS = full analysis set; PAS = primary analysis set; PK = pharmacokinetic.

#### 5. <u>STATISTICAL ANALYSES</u>

The analyses described in this SAP will supersede those specified in Protocol YO42373 for the purposes of a regulatory filing.

#### 5.1 GENERAL CONSIDERATION

All efficacy analyses will be performed on the PAS and the full analysis set (FAS), unless otherwise specified. Patients will be analyzed according to the treatment assigned at randomization by IxRS, regardless of whether they receive any assigned study drug.

Safety analyses will be conducted on the safety evaluable set, and will be performed based on the actual treatment patients received. Specifically, a patient will be included in the Tira+ACE arm in the safety analyses if the patient receives any amount of tiragolumab, regardless of the initial treatment assignment at randomization.

Unless otherwise stated, baseline values are the last available data obtained prior to the patient receiving the first dose of study treatment on Cycle 1, Day 1 (or at screening, for patients who were not treated).

#### 5.2 PATIENT DISPOSITION

Study enrollment and reasons for discontinuation from the study will be summarized by treatment arm for the FAS. Study treatment disposition and reasons for discontinuation from study treatment will be summarized for the safety evaluable set.

#### 5.3 PRIMARY ENDPOINTS ANALYSIS

# 5.3.1 <u>Definition of Co-Primary Endpoints</u>

The co-primary efficacy endpoints are PFS as assessed by the investigator according to RECIST v1.1 and OS in the PAS.

#### 5.3.1.1 Progression-Free Survival

The estimand is defined as follows:

- <u>Population</u>: Patients with previously untreated extensive-stage small cell lung cancer without presence or history of brain metastases at baseline
- <u>Variable</u>: Time from randomization to the first documented disease progression as determined by the investigator with the use of RECIST v1.1 or death from any cause, whichever occurs first.

#### Treatments:

- Experimental: tiragolumab+atezolizumab+CE (induction phase; four 21-day cycles) followed by tiragolumab+atezolizumab (maintenance phase; 21-day cycles)
- Control: placebo+atezolizumab+CE (induction phase; four 21-day cycles)
   followed by placebo+atezolizumab (maintenance phase; 21-day cycles)

#### Intercurrent events:

- Start of non-protocol anti-cancer therapy (NPT) prior to a PFS event
- Early discontinuation from study treatment for any reason prior to a PFS event
- Handling of intercurrent events: A treatment-policy with regards to the intercurrent events listed above will be applied for the primary analysis of PFS
- Summary measure: HR for PFS

Patients who have not experienced disease progression and have not died by the data cutoff date will be censored at the date of the last tumor assessment. Patients with no post-baseline tumor assessment will be censored at the date of randomization

#### 5.3.1.2 Overall Survival

The estimand is defined as the follows:

- <u>Population</u>: Patients with previously untreated extensive-stage small cell lung cancer without presence or history of brain metastases at baseline
- Variable: Time from randomization to death from any cause
- Treatments:
  - Experimental: tiragolumab+ atezolizumab+ CE (induction phase; four 21-day cycles) followed by tiragolumab+ atezolizumab (maintenance phase; 21-day cycles)
  - Control: placebo+ atezolizumab+ CE (induction phase; four 21-day cycles) followed by placebo+ atezolizumab (maintenance phase; 21-day cycles)

#### Intercurrent events:

- Start of NPT
- Early discontinuation from study treatment for any reason
- Handling of intercurrent events: A treatment-policy with regards to the intercurrent events listed above will be applied for the primary analysis of OS
- Summary measure: Hazard ratio for OS

Patients who are not reported as having died by the data cutoff date will be censored at the date when they were last known to be alive. Patients with no post-baseline information will be censored at the date of randomization.

# 5.3.2 Main Analytical Approach for Primary Endpoints



# 5.3.3 Handling of Missing Data

Patients who are lost to follow-up will be censored at the last date they were known to be alive for the primary analysis of OS. If > 5% of patients are lost to follow-up for OS in either treatment arm, a sensitivity analysis will be performed for the comparisons between two treatment arms in which patients who are lost to follow-up will be considered as having died at the last date they were known to be alive.

# 5.3.4 <u>Sensitivity Analyses for Primary Endpoints</u>

Sensitivity analyses of the primary endpoints will be performed to assess the impact of stratification. These analyses will follow the same analyses method as the primary endpoints with the exception that PFS and OS will be compared using a stratified log-rank test and the HR will be estimated from stratified Cox regression hazard model according to the protocol-defined stratification factors as entered in IxRS for the PAS (see also Section 5.3.2).

When the clinical effect is delayed by >20% of the median OS of the control group, a sensitivity analysis of OS may be performed using the weighted log-rank test based on the Rho-Gamma weight function family (Fleming and Harrington, 1991) or piece-wise linear weight functions (Lin and Leon, 2017) that weight more heavily on late events to account for the delayed clinical effect (Fine, 2007). In addition, hazard ratio estimates based on the corresponding Cox model (Lin and Leon, 2017) using the piece-wise linear weight functions may also be provided to enhance clinical interpretation of the treatment effect that varies over time.

# 5.3.5 <u>Supplementary Analyses for Primary Endpoints</u>

The following supplementary analyses will be performed for the co-primary efficacy endpoints of PFS and OS in which a different handling rule of intercurrent events is implemented to provide further understanding of the treatment effect.

#### 5.3.5.1 Subgroup Analyses for Primary Endpoints

The generalizability of OS and PFS results when comparing the Tira+ACE arm to the Pbo+ACE arm will be investigated by estimating the treatment effect in subgroups defined by demographics (e.g., age, sex) and baseline prognostic characteristics (e.g.,

ECOG Performance Status, LDH). Summaries of OS and PFS, including unstratified HRs estimated from Cox proportional hazards models and Kaplan-Meier estimates of median PFS and OS will be provided separately for each level of the subgroups for the comparisons between treatment arms.

#### 5.4 SECONDARY ENDPOINTS ANALYSES

# 5.4.1 Key Secondary Endpoints

# 5.4.1.1 Progression-Free Survival and Overall Survival in the Full Analysis Set

The estimand is defined similarly as for the co-primary endpoints of PFS and OS in Section 5.3.1 with the exception of the following:

Population: Patients with previously untreated extensive-stage small cell lung cancer.

Same analytical approaches for primary analysis of PFS and OS specified in Section 5.3 will be used to analyze PFS and OS on the FAS.

Subgroup analyses of PFS and OS on the FAS will also be provided by the baseline prognostic factor of presence or history of brain metastases.

### 5.4.1.2 Confirmed Overall Response Rate

The estimand for confirmed overall response rate (ORR) is defined as follows:

- <u>Population</u>: Patients with previously untreated extensive-stage small cell lung cancer without presence or history of brain metastases at baseline
- <u>Variable</u>: Whether patients achieved a confirmed objective response (i.e., complete response [CR] or partial response [PR] on two consecutive occasions ≥4 weeks apart), as determined by the investigator according to RECIST v1.1

#### Treatments:

- Experimental: tiragolumab+atezolizumab+CE (induction phase; four 21-day cycles) followed by tiragolumab+atezolizumab (maintenance phase; 21-day cycles)
- Control: placebo + atezolizumab + CE (induction phase; four 21-day cycles)
   followed by placebo + atezolizumab (maintenance phase; 21-day cycles)

#### Intercurrent events:

- Start of non-protocol anti-cancer therapy prior to a confirmed objective response is observed
- Early discontinuation from study treatment for any reason prior to a confirmed objective response is observed
- Handling of intercurrent events: a treatment-policy with regards to the intercurrent events listed above will be applied
- Summary measure: difference in proportions of patients achieved confirmed objective response between treatments

An alternative estimand for confirmed ORR is defined similarly as above with the exception of the following:

<u>Population</u>: patients with previously untreated extensive-stage small cell lung cancer

Confirmed ORR will be analyzed in patients with measurable disease at baseline and compared between treatment arms using Chi-square test. The 95% CI for the difference in confirmed ORRs between the two treatment arms will be computed using the Newcombe method. The 95% CI of the confirmed ORR will be calculated for each treatment arm using the Wilson score method.

# 5.4.2 Supportive Secondary Endpoint(s)

# 5.4.2.1 **Duration of Response**

Duration of response (DOR) will be assessed in the PAS and the FAS for patients who achieved a confirmed objective response, as determined by the investigator according to RECIST v1.1. DOR is defined as time from the date of the first occurrence of a confirmed objective response until the first date of progressive disease as determined by the investigator according to RECIST v1.1 or death from any cause, whichever occurs first. Patients who have not progressed and who have not died at the time of analysis will be censored at the time of the last tumor assessment date. DOR will be based on a non-randomized subset of patients (specifically, patients who achieve a confirmed objective response); therefore, hypothesis testing will not be performed for this endpoint. Comparisons between treatment arms will be made for descriptive purposes. Median DOR and corresponding 95% CIs will be estimated using Kaplan-Meier methodology for each treatment arm.

#### 5.4.2.2 PFS and OS Rates at Selected Time Points

The PFS rates at 6 months and at 12 months are defined as the proportion of patients who have not experienced disease progression as determined by the investigator according to RECIST v1.1 or death from any cause at 6 months and 12 months after randomization. The PFS rates will be estimated using Kaplan-Meier methodology for each treatment arm, along with 95% CIs calculated using the standard error derived from Greenwood's formula. The 95% CI for the difference in PFS rates between the two treatment arms will be estimated using the normal approximation method, with standard errors computed using Greenwood's method.

Similar analyses will be performed for the OS rates at 1 and 2 years, defined as the proportion of patients who have not died from any cause at 12 months and 24 months after randomization.

# 5.4.2.3 Time to Confirmed Deterioration in Physical Functioning and Global Health Status

Patient-reported physical functioning (items 1-5) and global health status (GHS)/ quality of life (QoL) (items 29-30) as collected and measured by the European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30

(QLQ-C30). A high score for the physical function subscale represents a high/healthy level of functioning and a high score for the GHS/QoL subscale represents a high health related quality of life. Both scales will be linearly transformed so that each score will range from 0 to 100. A score change of at least 10-point in GHS/QoL and functional subscale score is perceived by patients as clinically meaningful (Osoba et al. 1998).

The estimand for time to confirmed deterioration (TTCD) is defined as the follows:

- <u>Population</u>: patients with previously untreated extensive-stage small cell lung cancer without presence or history of brain metastases at baseline
- <u>Variable</u>: Time from randomization until the first confirmed clinically meaningful
  deterioration on physical functioning and GHS/QoL EORTC QLQ-C30 select scales;
  confirmed clinically meaningful deterioration is defined as a clinically meaningful
  decrease from baseline that must be held for at least two consecutive assessments
  or an initial clinically meaningful decrease from baseline followed by death from any
  cause within 3 weeks.

#### Treatments:

- Experimental: tiragolumab+atezolizumab+CE (induction phase; four 21-day cycles) followed by tiragolumab+atezolizumab (maintenance phase; 21-day cycles)
- Control: placebo+atezolizumab+CE (induction phase; four 21-day cycles)
   followed by placebo+atezolizumab (maintenance phase; 21-day cycles)
- Intercurrent events:
  - Start of NPT prior to a confirmed clinical meaningful deterioration
  - Early discontinuation from study treatment for any reason prior to a confirmed clinical meaningful deterioration
  - Death that occurs before patients report any clinically meaningful deterioration
- Handling of intercurrent events: A treatment policy strategy with regards to the start
  of NPT and early discontinuation; and while-on-treatment/while-alive strategy for
  death will be applied for the TTCD analysis.
- Summary measure: Hazard Ratio for TTCD

An alternative estimand for TTCD is defined similarly as above with the exception of the following:

Population: patients with previously untreated extensive-stage small cell lung cancer

For patients who discontinue study treatment for radiographic disease progression per RECIST v1.1 and enter the survival follow-up, the questionnaires will be completed at 3 months (±30 days) and 6 months (±30 days) following the visit in which progressive disease was confirmed. Patients who have not experienced a confirmed clinically meaningful deterioration by the clinical cutoff date will be censored at the last time when they completed an assessment. Patients with no baseline or post-baseline assessment will be censored at the date of randomization. According to the while on treatment/while-

alive strategy, patients who died before reporting any clinical meaningful deterioration will be censored at the last time when they completed an assessment. TTCD will be analyzed using the same methods as for the co-primary endpoint of PFS.

# 5.5 EXPLORATORY ENDPOINTS ANALYSIS

# 5.5.1 <u>Patient Reported Outcomes</u>



#### 5.6 SAFETY ANALYSES

Unless specified otherwise, safety analyses described below will be conducted for the safety evaluable set (see Section 5.4), with participants grouped according to whether any tiragolumab was received.

# 5.6.1 <u>Extent of Exposure</u>

Study drug exposure, including treatment duration, dosage, and dose intensity, will be summarized by treatment arm and for each study drug with descriptive statistics.

#### 5.6.2 Adverse Events

Verbatim description of AEs will be mapped to the Medical Dictionary for Regulatory Activities (MedDRA) thesaurus terms. Severity for all adverse events will be graded by the investigator according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0, and severity for cytokine-release syndrome (CRS) will also be graded by the investigator according to the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading scale.

All treatment-emergent adverse events will be summarized by treatment arm and NCI CTCAE grade. CRS will also be summarized by treatment arm and the ASTCT consensus grade. In addition, common adverse events, treatment-related AEs, serious adverse events (SAEs), adverse events leading to study treatment discontinuation or interruption, Grade 3-4 AEs, and fatal AE (Grade 5) will be summarized accordingly. For the purpose of analyses, adverse events of special interest (AESI) are identified by a set of comprehensive definitions using standardized MedDRA queries (SMQs), High-Level Terms (HLTs) and Sponsor-defined adverse event grouped terms (AEGTs) from the AE clinical database by medical concept. The AESI will be summarized by treatment arm and CTCAE grade.

Multiple occurrence of the same event will be counted once at the maximum severity.

For the safety analyses, "treatment-emergent" is defined as adverse events occurring on or after the first dose of study drug treatment or pre-existing condition that worsened on or after the first dose of the study treatment up to the data cutoff date.

Key adverse events that occurred during the induction and maintenance therapy phases may also be summarized separately.

Listings of adverse events will include all treatment emergent adverse events up to the data cutoff date.

Deaths during the study treatment period and those reported during the follow-up period after treatment completion or discontinuation and causes of death will be summarized by treatment arm.

## 5.6.3 Laboratory Data

Laboratory data will be summarized by treatment arm. Selected laboratory data will be graded according to NCI CTCAE v5.0 and will be summarized descriptively. Shift tables from baseline to worst post-baseline values will also be presented.

## 5.6.4 <u>Vital Signs</u>

Vital signs will be summarized by treatment arm and visit.

#### 5.7 OTHER ANALYSES

## 5.7.1 Summaries of Conduct of Study

Study enrollment and major protocol deviations including major deviations of inclusion/exclusion criteria will be summarized by treatment arm for the FAS.

# 5.7.2 <u>Summaries of Treatment Group Comparability</u>

Demographic characteristics (e.g., as age, sex), baseline prognostic characteristics (e.g., smoking status) and stratification factors (ECOG Performance Status, LDH) will be summarized by treatment arm for the FAS and the PAS.

Descriptive statistics (mean, median, standard deviation, and range) will be presented for continuous variables, and frequencies and percentages will be presented for categorical variables.

#### 5.7.3 Pharmacokinetic Analyses

Serum concentrations of tiragolumab and atezolizumab will be reported as individual values and summarized (mean, standard deviation, coefficient of variation, median, range, geometric mean, and geometric mean coefficient of variation) by treatment arm and cycle, when appropriate and as data allow. Individual and median serum tiragolumab and atezolizumab concentrations will be plotted by treatment arm and day.

Additional PK analyses may be conducted, as appropriate, based on the availability of data.

All PK analyses will be conducted on the PK-evaluable set.

#### 5.7.4 Immunogenicity Analyses

The immunogenicity analyses will include patients with any tiragolumab anti-drug antibody (ADA) assessments, with patients grouped according to the treatment received.

The number and proportion of treatment-emergent tiragolumab ADA-positive patients will be summarized for the Tira+ACE arm..

Demographic and baseline characteristics, PK, efficacy, and safety by treatmentemergent tiragolumab ADA subgroups may be reported.

Immunogenicity analyses will be conducted on the tiragolumab ADA-evaluable sets.

#### 5.8 INTERIM ANALYSES

## 5.8.1 Planned Interim Analyses

There are no planned interim analyses of the co-primary endpoint of PFS and OS.

# 6. SUPPORTING DOCUMENTATION

This section is not applicable, since there is no additional supporting document.

### 7. <u>REFERENCES</u>

- Akazawa KO, Nakamura T, Palesch Y. Power of logrank test and Cox regression model in clinical trials with heterogeneous samples. Stat Med. 1997;16:583-97.
- Basch E, Reeve BB, Mitchell SA, et al. Development of the National Cancer Institute's patient-reported outcomes version of the common terminology criteria for adverse events (PRO-CTCAE). J Natl Cancer Inst 2014;106:1-11.
- Brookmeyer R, Crowley J. A confidence interval for the median survival time. Biometrics 1982:38:29-41.
- Fine GD. Consequences of delayed treatment effects on analysis of time-to-event endpoints. Ther Innov Regul Sci 2007;41:535–9.
- Fleming TR, Harrington DP. Counting processes and survival analysis. New York: John Wiley Sons, 1991.
- Lin RS, León LF. Estimation of treatment effects in weighted log-rank tests. Contemporary clinical trials communications. 2017;8:147-55.
- Osoba D, Rodrigues G, Myles J, et al. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol 1998;16:139–44.

# Signature Page for Statistical Analysis Plan - YO42373 -Published System identifier: RIM-CLIN-441594

| Approval Task | |
|---------------|-------------------------------|
| | Company Signatory |
| | 27-May-2022 13:27:57 GMT+0000 |